CLINICAL TRIAL: NCT02307409
Title: Assessment of Coagulation Profile and Haematopoietic Responses in Patients With Acute-on-chronic Liver Failure During Systemic Inflammatory Response (SIRS) and Sepsis
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-SIRS-01
Record Dates: First submitted 2014-11-18; First posted 2014-12-04 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2016-04

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Decompensated Chronic Liver Disease: Decompensated Chronic Liver Disease patients will be enrol
  Interventions: Other: Sonoclot/TEG test
- Healthy Controls: Healthy Controls will be enrol
  Interventions: Other: Sonoclot/TEG test

INTERVENTIONS:
Other: Sonoclot/TEG test — The Sonoclot/TEG test will be done at the study time points. Within 12 hours of presentation in the emergency department, at 72 hours, and at 7 days, or when the patient meets the study criteria for suspected or proven sepsis

SUMMARY:
This study attempts to clarify the pathophysiology of haemostasis and haematopoiesis in relation to the evidence of sepsis in liver disease, and compares the accuracy of various available laboratory tests in assessment of these patients. Further research is needed for proper understanding of the influence of sepsis on coagulation disorders in ACLF (Acute on Chronic Liver Failure) patients in particular, to correctly identify the type and optimal quantity of blood product requirement in at risk patients.

Thromboelastography (TEG) /Sonoclot have been proposed as a superior tool to rapidly diagnose and help guide resuscitation with blood products. Secondly, the study of derangement in coagulopathy after the onset of sepsis is of paramount importance because of increased mortality after the onset of sepsis. In the present study, patients with ACLF (Acute on Chronic Liver Failure) without evidence of sepsis on admission will be included in the study cohort, and will undergo a baseline diagnostic workup as described. They will be followed for development of any signs of infection after hospitalization. Then the effect of sepsis on their coagulation and haematopoietic cellular responses will be assessed. Thus the effect of sepsis on the progression and outcome of patients with ACLF (Acute on Chronic Liver Failure) will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* ACLF (Acute on Chronic Liver Failure), as diagnosed by APASL (Asian Pacific association of Study of Liver Disease) criteria mentioned above.

Exclusion Criteria:

* Patients with evidence of sepsis at presentation.
* Current therapy: Recent blood or blood component transfusion in the last 2 days.
* HIV positive/ AIDS patients
* Patients requiring anti platelet therapy,
* Renal insufficiency requiring dialysis
* Active malignancy within the last 5 years
* Patient with other neurological disease and metabolic disorders, unbalanced heart failure and/or respiratory failure or end-stage renal disease
* Administration of anticoagulants, antifibrinolytics,
* Not willing to participate in the study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population for this study is all Acute on Chronic Liver Failure patients admitted to the inpatient services of ILBS, New Delhi.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Prevalence and severity of coagulation profile derangement and haematopoietic responses, by sonoclot/ TEG, coagulation and hematological parameters, in acute- on-chronic liver failure with and without systemic inflammatory response. | 0 day, 3 day & 7 day after admission.

SECONDARY OUTCOMES:
Utility of sonoclot/ TEG in predicting blood product utilization. | 0 day, 3 day & 7 day after admission.
  Reporting of blood product usage in 7 days of admission as per TEG R time, K time, Maximum amplitude of curve, angle, lysis at 30%.
Sonoclot/TEG result indicating hypocoagulability correlates with the patient's tendency to bleed in ACLF. | 0 day, 3 day & 7 day after admission.
  Reporting of number and site of bleed- skin, mucosa, urine, GI tract, CNS etc.
Changes in baseline coagulation profile can predict development of sepsis in patients of ACLF. | 0 day, 3 day & 7 day after admission.
  Correlation of PT/INR with TEG parameters and positive blood or urine culture.
Coagulation dysfunction (prothrombotic and anticoagulant tendencies) in patients with ACLF with or without evidence of sepsis. | 0 day, 3 day & 7 day after admission.
Effect of sepsis on the haematopoietic response of patients with Acute on Chronic Liver Failure. | 0 day, 3 day & 7 day after admission.
  Measurement of reticulocyte count, and peripheral amear- presence of toxic granules.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Premkumar M, Bihari C, Saxena P, Devurgowda DR, Vyas T, Mirza R, Jain P, Kumar G, Bhatia P, Baweja S, Choudhury A, Sarin SK. Heparin-like Effect Associated With Risk of Bleeding, Sepsis, and Death in Patients With Severe Alcohol-Associated Hepatitis. Clin Gastroenterol Hepatol. 2020 Feb;18(2):486-495.e3. doi: 10.1016/j.cgh.2019.04.057. Epub 2019 May 8. PMID 31077821
- [Derived] Premkumar M, Saxena P, Rangegowda D, Baweja S, Mirza R, Jain P, Bhatia P, Kumar G, Bihari C, Kalal C, Vyas T, Choudhury A, Sarin SK. Coagulation failure is associated with bleeding events and clinical outcome during systemic inflammatory response and sepsis in acute-on-chronic liver failure: An observational cohort study. Liver Int. 2019 Apr;39(4):694-704. doi: 10.1111/liv.14034. Epub 2019 Feb 7. PMID 30589495